CLINICAL TRIAL: NCT07182331
Title: Effects of cTBS on Sensory Integration in Children With Autism Spectrum Disorder: A Randomized, Sham-Controlled Study Integrating Genetic Markers, MRI, fNIRS, and Temporal Binding Tasks
Brief Title: Brain Stimulation and Sensory Integration in Children With ASD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Neurolab Plus (Industry)
Collaborators: Al-Farabi Kazakh National University (KazNU) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2.2.6.1; BR27198099 (Other Grant/Funding Number: Non-profit joint-stock company "Al-Farabi Kazakh National University")
Record Dates: First submitted 2025-08-20; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: Transcranial Magnetic Stimulation; Theta Burst Stimulation; Pediatric Neurostimulation; Neurodevelopmental Disorders; Multimodal Biomarkers; Electrophysiology; Functional Near-Infrared Spectroscopy; Magnetic Resonance Imaging; Genetic Markers; Randomized Controlled Trial; Sham-Controlled Trial; Child Neuropsychology; Autism Spectrum Disorder; Sensory Processing; Audiovisual Integration; Temporal Binding Window; Sound-Induced Flash Illusion; Temporal Perception
MeSH Terms: conditions — Autism Spectrum Disorder; Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, investigators, and outcome assessors are all blinded to group assignment (active vs. sham TMS). The sham condition mimics the sound and sensation of stimulation without delivering active magnetic pulses, using an identical setup. Randomization and group codes are maintained by an independent administrator and not revealed until after final data analysis. Blinding is used to reduce bias in behavioral, neurophysiological, and questionnaire-based outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active cTBS to Bilateral DLPFC (Experimental): Participants receive active continuous theta burst stimulation (cTBS) targeting both the left and right dorsolateral prefrontal cortex (DLPFC) during each session. Stimulation is delivered consecutively to both hemispheres using a standard cTBS protocol: 600 pulses per side (triplet bursts at 50 Hz, repeated at 5 Hz), with each hemisphere receiving stimulation over approximately 40 seconds, at 80% of the individual's active motor threshold. A total of 10 bilateral sessions are delivered over two weeks.
  Interventions: Device: Continuous Theta Burst Stimulation to Bilateral DLPFC
- Sham cTBS to Bilateral DLPFC (Sham Comparator): Participants receive sham stimulation to both the left and right DLPFC during each session. Procedures mimic the active condition, including coil placement, session duration, and auditory cues, but no effective magnetic pulses are delivered. Each participant completes 10 bilateral sham sessions over two weeks. The protocol maintains blinding to control for placebo effects and procedural expectations.
  Interventions: Device: Sham Continuous Theta Burst Stimulation

INTERVENTIONS:
Device: Continuous Theta Burst Stimulation to Bilateral DLPFC — Participants receive continuous theta burst stimulation (cTBS) targeting both the left and right dorsolateral prefrontal cortex (DLPFC) during each session. Each hemisphere is stimulated with 600 pulses (triplets at 50 Hz repeated at 5 Hz) over ~40 seconds, at 80% of the individual's active motor threshold. Sessions are administered once daily over 10 treatment days.
  Other Names: cTBS
  Arms: Active cTBS to Bilateral DLPFC
Device: Sham Continuous Theta Burst Stimulation — Participants receive sham continuous theta burst stimulation (cTBS) to both the left and right dorsolateral prefrontal cortex (DLPFC) using a placebo coil that mimics the auditory and tactile sensations of real stimulation but does not produce a magnetic field capable of affecting brain activity. Coil positioning, session timing, and procedure match the active cTBS protocol, including consecutive stimulation to both hemispheres. Both participants and TMS technicians wear earplugs to mask subtle sound differences between active and sham coils. This setup maintains participant and operator blinding and controls for placebo-related effects.
  Other Names: Sham cTBS
  Arms: Sham cTBS to Bilateral DLPFC

SUMMARY:
The goal of this clinical trial is to find out if brain stimulation can help improve sensory integration in children ages 6 to 12 with autism spectrum disorder (ASD). The main questions it aims to answer are:

Does brain stimulation using continuous theta-burst stimulation (cTBS) on bilateral dorsolateral prefrontal cortex (DLPFC) improve how children process sights and sounds together? Can brain functioning, structure, and genetics help predict who responds best to this treatment?

Researchers will compare the results of the randomly assigned active brain stimulation to sham (inactive) stimulation groups to see if the treatment works.

Participants will:

Receive 10 sessions of either active or sham cTBS over 2 weeks Complete a sensory task involving flashes and beeps before and after stimulation Take part in brain scans, namely magnetic resonance imaging (MRI) and functional near-infrared spectroscopy (fNIRS), and provide a saliva sample for genetic testing

DETAILED DESCRIPTION:
This study explores how noninvasive brain stimulation may support children with Autism Spectrum Disorder (ASD) by improving how their brains process and combine sounds and images. It also investigates whether changes in brain function, brain structure, and specific genes can help predict how well a child might respond to this type of stimulation. The study is focused on a core challenge in ASD: differences in how children experience sensory input-especially how their brains process what they see and hear together.

The central concept in this research is something called the Temporal Binding Window (TBW). TBW refers to the brief time window in which the brain naturally fuses sensory information from different senses-like sight and sound-into a single event. For most people, this window is quite narrow: sounds and images that are even slightly out of sync are perceived as separate. But in many children with ASD, this window is wider. That means they may confuse the order or timing of sensory inputs, which can affect communication, behavior, and learning.

To address this, the study uses a method called transcranial magnetic stimulation (TMS). This technique delivers brief, painless pulses of magnetic energy to the surface of the brain using a special coil held against the scalp. The type of TMS used here is called continuous theta burst stimulation (cTBS), which delivers rapid bursts of magnetic pulses designed to gently decrease the excitability of targeted brain areas. In this study, cTBS is used to modulate activity in a region called the dorsolateral prefrontal cortex (DLPFC), which is important for regulating attention, working memory, and sensory control.

A total of 40 children between the ages of 6 and 12 will take part. All participants must have a formal diagnosis of ASD, confirmed using a structured caregiver interview known as the Autism Diagnostic Interview - Revised (ADI-R). They must also demonstrate average or above-average cognitive ability, based on a two-subscale IQ measure from the Wechsler Intelligence Scale for Children - Fifth Edition (WISC-V). This ensures that all children can understand the tasks and safely undergo the procedures.

Participants are randomly assigned to one of two groups: an active TMS group or a sham TMS group. In the sham group, the same equipment is used, but no actual magnetic stimulation reaches the brain. This allows researchers to compare outcomes while keeping the children, their families, and the staff unaware of group assignments.

Each child completes ten sessions of either active or sham TMS, over approximately two weeks. The stimulation is applied alternately to the left and right sides of the forehead area, corresponding to the DLPFC. Each session lasts only a few minutes. The stimulation is calibrated individually using a simple test to determine the strength needed to trigger a small movement in the child's hand. All children wear ear protection and are supervised closely by trained staff.

The main outcome of the study is a measure of how well children can process timing between visual and auditory signals. This is assessed using a behavioral task known as the Sound-Induced Flash Illusion (SIFI). In this task, the child looks at a screen and hears beeps while seeing flashes of light. Sometimes there is only one flash, but if it is paired with two quick beeps, some children perceive two flashes instead of one. By changing the timing between the flash and the beeps, researchers can measure the range of delays where the child still experiences the illusion. This range is called the Temporal Binding Window. The wider the window, the more likely the child's brain is to "fuse" signals that actually happened at different times. This task is performed before and after the TMS intervention.

In addition to this behavioral task, the study uses two caregiver questionnaires to track any changes in symptoms:

The Autism Treatment Evaluation Checklist (ATEC) is a brief form filled out by parents. It includes four sections: communication skills, social behavior, sensory awareness, and physical health. It is used to detect broad changes in behavior and well-being.

The Short Sensory Profile (SSP) is another caregiver questionnaire that focuses on how children respond to sensory experiences. It includes questions about sensitivity to touch, sound, movement, and visual stimuli.

These tools are chosen because they are simple, validated, and commonly used in ASD research. They are also sensitive to changes in daily functioning and sensory behavior.

To explore how brain function might change as a result of stimulation, the study uses a technique called functional near-infrared spectroscopy (fNIRS). This is a safe, quiet, and noninvasive method that measures how much oxygen is in the blood within specific brain regions. The child wears a soft cap with small sensors that shine near-infrared light into the scalp. This light reflects back differently depending on how much oxygen is being used in the brain underneath. The sensors are placed over the same area that receives the stimulation (the prefrontal cortex), and the recording is done while the child sits quietly with eyes open. There is no task or performance required-this is simply a measurement of the brain's resting state. Recordings are done once before the stimulation begins and again after the final session.

The study also includes a one-time brain scan using magnetic resonance imaging (MRI). MRI provides a detailed image of the structure of the brain, including its size, shape, and thickness in different regions. This helps researchers look for any physical brain characteristics that might explain differences in sensory processing or predict whether a child will respond to the stimulation. The scan is done in a hospital or imaging center using standard pediatric procedures. Children are given headphones, padding, and visual aids to help them feel comfortable and reduce movement. They do not receive any injections or medications.

Finally, the study includes a one-time saliva collection to analyze DNA. This is done using a small sterile tube into which the child spits or where saliva is collected using a swab. The sample is stored and later processed in a genetics lab. Researchers analyze specific single-nucleotide polymorphisms in genes known to be involved in brain development and sensory processing. These include genes such as SHANK3, CNTNAP2, NRXN1, and SCN2A. The goal is to determine whether certain gene variants are associated with differences in how children respond to the stimulation or process multisensory information. This part of the study is exploratory and does not involve returning results to families.

All procedures are conducted in compliance with safety guidelines for pediatric brain stimulation and neuroimaging. Children are monitored throughout the study, and staff are trained to recognize and manage any discomfort or side effects. The TMS procedures are designed to be brief, well-tolerated, and minimally invasive. Participation is voluntary, and families can withdraw at any time.

This research is part of a broader effort to develop personalized approaches to brain stimulation in children with developmental conditions. By combining behavioral tasks, brain imaging, and genetics, the study aims to understand which children are most likely to benefit from neuromodulation and how their sensory systems can be supported. The long-term goal is to inform clinical interventions that are evidence-based, child-centered, and tailored to individual needs.

This study is conducted at a research site in Almaty, Kazakhstan and is funded by the Ministry of Science and Higher Education of the Republic of Kazakhstan under grant number IRN BR27198099. Ethical approval was obtained from the Local Ethical Committee of Al-Farabi Kazakh National University (Protocol No. IRB-A843). The study does not involve U.S. FDA-regulated products and is not conducted under an IND or IDE.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-12 years at the time of enrollment.
* Clinical diagnosis of Autism Spectrum Disorder (ASD) confirmed using the Autism Diagnostic Interview-Revised (ADI-R).
* Intelligence quotient (IQ) ≥ 70 as measured by the General Ability Index (GAI) from the Wechsler Intelligence Scale for Children - Fifth Edition (WISC-V).
* Ability to understand and follow simple instructions for behavioral tasks and stimulation procedures.
* Stable medication regimen (if any) for at least 4 weeks before the start of the study.
* Written informed consent from a parent or legal guardian, and assent from the child when appropriate.

Exclusion Criteria:

* History of epilepsy, seizures, or abnormal EEG suggestive of seizure risk.
* Presence of metal implants, devices, or foreign bodies in or near the head (except dental fillings) that are contraindicated for TMS or MRI.
* Serious neurological disorders other than ASD (e.g., cerebral palsy, brain injury, neurodegenerative disease).
* Severe psychiatric disorders requiring hospitalization or urgent intervention.
* Current or past history of significant head trauma with loss of consciousness > 5 minutes.
* Uncorrected hearing or vision problems that could interfere with task performance.
* Inability to tolerate sitting still for 15-20 minutes.
* Participation in another interventional clinical trial within the past 3 months.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Temporal Binding Window (TBW) Width Measured Using the Sound-Induced Flash Illusion (SIFI) Task | Baseline and up to 7 days after the final TMS session.
  The TBW reflects the time interval within which auditory and visual stimuli are integrated as a single percept. It is assessed by computing the proportion of illusion-consistent responses across varying stimulus onset asynchronies in the SIFI task. A reduction in TBW width, measured in milliseconds (ms) following stimulation indicates improved multisensory temporal precision.

SECONDARY OUTCOMES:
Change in Sensory Processing Profile (Short Sensory Profile, SSP) | Baseline and up to 7 days after the final TMS session.
  Parent-reported Short Sensory Profile (SSP; total score range: 38-190). Lower scores indicate greater difficulties with sensory processing. Changes in total and subscale scores will be reported.
Change in Autism Symptom Severity (Autism Treatment Evaluation Checklist, ATEC) | Baseline and up to 7 days after the final TMS session.
  Parent-reported Autism Treatment Evaluation Checklist (ATEC; total score range: 0-179). Higher scores indicate greater severity. Subscales include communication, sociability, sensory/cognitive awareness, and health/physical behavior.
Change in Resting-State Prefrontal Activity - Mean Oxygenation (fNIRS) | Baseline and up to 7 days after the final TMS session.
  Description: Resting-state functional near-infrared spectroscopy (fNIRS) measurement of mean oxygenated hemoglobin (HbO, µM) in the dorsolateral prefrontal cortex (DLPFC).
Change in Resting-State Prefrontal Activity - Functional Connectivity (fNIRS) | Baseline and up to 7 days after the final TMS session.
  Resting-state fNIRS measurement of connectivity indices across DLPFC channels (e.g., correlation coefficients between HbO time series).

OTHER OUTCOMES:
Correlation of Cortical Thickness (MRI) with Change in TBW Width (SIFI) | MRI obtained once at baseline.
  Cortical thickness (mm) in prefrontal, temporal, and sensory-integration regions measured with structural MRI at baseline will be correlated with change in Temporal Binding Window (TBW) width (ms) from the Sound-Induced Flash Illusion task.
Correlation of Cortical Volume (MRI) with Change in TBW Width (SIFI) | MRI obtained once at baseline.
  Cortical volume (mm³) in prefrontal, temporal, and sensory-integration regions measured with structural MRI at baseline will be correlated with the change in TBW width (ms).
Correlation of Genetic Variant Frequencies with Change in TBW Width (SIFI) | Saliva samples collected once at baseline.
  Frequencies of alleles/genotypes for pre-specified single-nucleotide polymorphisms (SNPs) associated with higher ASD risk or symptom severity obtained from saliva DNA and correlated with change in TBW width (ms).

CONTACTS AND LOCATIONS:
Locations (2):
- Kazakhstan (2):
  - Neurolab Plus, Almaty
  - Non-profit joint-stock company "Al-Farabi Kazakh National University", Almaty

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including demographics, baseline and outcome measures from the Sound-Induced Flash Illusion (SIFI) task, Autism Treatment Evaluation Checklist (ATEC), Short Sensory Profile (SSP), genetic markers (saliva DNA sequencing results limited to specified polymorphisms), structural MRI volumetric data, fNIRS prefrontal oxygenation measures, and TMS stimulation parameters, will be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: De-identified data will be made available within 12 months following publication of the main study results and will remain available for at least 5 years thereafter.
Access Criteria: Data will be accessible to qualified researchers at academic or medical institutions upon submission of a justified request. Each request will be reviewed by the study steering committee. Approved researchers will sign a data use agreement to ensure compliance with ethical standards, including prohibiting any attempt to re-identify participants. Data will be distributed via a secure repository.
URL: https://osf.io/mz79u

REFERENCES:
- [Background] Siemann JK, Veenstra-VanderWeele J, Wallace MT. Approaches to Understanding Multisensory Dysfunction in Autism Spectrum Disorder. Autism Res. 2020 Sep;13(9):1430-1449. doi: 10.1002/aur.2375. Epub 2020 Sep 1. PMID 32869933
- [Background] Wallace MT, Stevenson RA. The construct of the multisensory temporal binding window and its dysregulation in developmental disabilities. Neuropsychologia. 2014 Nov;64:105-23. doi: 10.1016/j.neuropsychologia.2014.08.005. Epub 2014 Aug 13. PMID 25128432
- [Background] Qiu S, Qiu Y, Li Y, Cong X. Genetics of autism spectrum disorder: an umbrella review of systematic reviews and meta-analyses. Transl Psychiatry. 2022 Jun 15;12(1):249. doi: 10.1038/s41398-022-02009-6. PMID 35705542
- [Background] Camasio A, Panzeri E, Mancuso L, Costa T, Manuello J, Ferraro M, Duca S, Cauda F, Liloia D. Linking neuroanatomical abnormalities in autism spectrum disorder with gene expression of candidate ASD genes: A meta-analytic and network-oriented approach. PLoS One. 2022 Nov 28;17(11):e0277466. doi: 10.1371/journal.pone.0277466. eCollection 2022. PMID 36441779
- [Background] Wang H, Ma ZH, Xu LZ, Yang L, Ji ZZ, Tang XZ, Liu JR, Li X, Cao QJ, Liu J. Developmental brain structural atypicalities in autism: a voxel-based morphometry analysis. Child Adolesc Psychiatry Ment Health. 2022 Jan 31;16(1):7. doi: 10.1186/s13034-022-00443-4. PMID 35101065
- [Background] Sokhadze EM, Lamina EV, Casanova EL, Kelly DP, Opris I, Tasman A, Casanova MF. Exploratory Study of rTMS Neuromodulation Effects on Electrocortical Functional Measures of Performance in an Oddball Test and Behavioral Symptoms in Autism. Front Syst Neurosci. 2018 May 28;12:20. doi: 10.3389/fnsys.2018.00020. eCollection 2018. PMID 29892214
- [Background] Casanova MF, Sokhadze EM, Casanova EL, Opris I, Abujadi C, Marcolin MA, Li X. Translational Neuroscience in Autism: From Neuropathology to Transcranial Magnetic Stimulation Therapies. Psychiatr Clin North Am. 2020 Jun;43(2):229-248. doi: 10.1016/j.psc.2020.02.004. Epub 2020 Apr 8. PMID 32439019
- [Background] Foss-Feig JH, Kwakye LD, Cascio CJ, Burnette CP, Kadivar H, Stone WL, Wallace MT. An extended multisensory temporal binding window in autism spectrum disorders. Exp Brain Res. 2010 Jun;203(2):381-9. doi: 10.1007/s00221-010-2240-4. PMID 20390256
- [Background] Hardan AY, Libove RA, Keshavan MS, Melhem NM, Minshew NJ. A preliminary longitudinal magnetic resonance imaging study of brain volume and cortical thickness in autism. Biol Psychiatry. 2009 Aug 15;66(4):320-6. doi: 10.1016/j.biopsych.2009.04.024. Epub 2009 Jun 11. PMID 19520362
- [Background] Grove J, Ripke S, Als TD, Mattheisen M, Walters RK, Won H, Pallesen J, Agerbo E, Andreassen OA, Anney R, Awashti S, Belliveau R, Bettella F, Buxbaum JD, Bybjerg-Grauholm J, Baekvad-Hansen M, Cerrato F, Chambert K, Christensen JH, Churchhouse C, Dellenvall K, Demontis D, De Rubeis S, Devlin B, Djurovic S, Dumont AL, Goldstein JI, Hansen CS, Hauberg ME, Hollegaard MV, Hope S, Howrigan DP, Huang H, Hultman CM, Klei L, Maller J, Martin J, Martin AR, Moran JL, Nyegaard M, Naerland T, Palmer DS, Palotie A, Pedersen CB, Pedersen MG, dPoterba T, Poulsen JB, Pourcain BS, Qvist P, Rehnstrom K, Reichenberg A, Reichert J, Robinson EB, Roeder K, Roussos P, Saemundsen E, Sandin S, Satterstrom FK, Davey Smith G, Stefansson H, Steinberg S, Stevens CR, Sullivan PF, Turley P, Walters GB, Xu X; Autism Spectrum Disorder Working Group of the Psychiatric Genomics Consortium; BUPGEN; Major Depressive Disorder Working Group of the Psychiatric Genomics Consortium; 23andMe Research Team; Stefansson K, Geschwind DH, Nordentoft M, Hougaard DM, Werge T, Mors O, Mortensen PB, Neale BM, Daly MJ, Borglum AD. Identification of common genetic risk variants for autism spectrum disorder. Nat Genet. 2019 Mar;51(3):431-444. doi: 10.1038/s41588-019-0344-8. Epub 2019 Feb 25. PMID 30804558
- [Background] Gavin N, Hirst RJ, McGovern DP. The magnitude of the sound-induced flash illusion does not increase monotonically as a function of visual stimulus eccentricity. Atten Percept Psychophys. 2022 Jul;84(5):1689-1698. doi: 10.3758/s13414-022-02493-4. Epub 2022 May 13. PMID 35562629
- [Background] De Rubeis S, He X, Goldberg AP, Poultney CS, Samocha K, Cicek AE, Kou Y, Liu L, Fromer M, Walker S, Singh T, Klei L, Kosmicki J, Shih-Chen F, Aleksic B, Biscaldi M, Bolton PF, Brownfeld JM, Cai J, Campbell NG, Carracedo A, Chahrour MH, Chiocchetti AG, Coon H, Crawford EL, Curran SR, Dawson G, Duketis E, Fernandez BA, Gallagher L, Geller E, Guter SJ, Hill RS, Ionita-Laza J, Jimenz Gonzalez P, Kilpinen H, Klauck SM, Kolevzon A, Lee I, Lei I, Lei J, Lehtimaki T, Lin CF, Ma'ayan A, Marshall CR, McInnes AL, Neale B, Owen MJ, Ozaki N, Parellada M, Parr JR, Purcell S, Puura K, Rajagopalan D, Rehnstrom K, Reichenberg A, Sabo A, Sachse M, Sanders SJ, Schafer C, Schulte-Ruther M, Skuse D, Stevens C, Szatmari P, Tammimies K, Valladares O, Voran A, Li-San W, Weiss LA, Willsey AJ, Yu TW, Yuen RK; DDD Study; Homozygosity Mapping Collaborative for Autism; UK10K Consortium; Cook EH, Freitag CM, Gill M, Hultman CM, Lehner T, Palotie A, Schellenberg GD, Sklar P, State MW, Sutcliffe JS, Walsh CA, Scherer SW, Zwick ME, Barett JC, Cutler DJ, Roeder K, Devlin B, Daly MJ, Buxbaum JD. Synaptic, transcriptional and chromatin genes disrupted in autism. Nature. 2014 Nov 13;515(7526):209-15. doi: 10.1038/nature13772. Epub 2014 Oct 29. PMID 25363760
- [Background] Casanova MF, Sokhadze EM, Casanova EL, Li X. Transcranial Magnetic Stimulation in Autism Spectrum Disorders: Neuropathological Underpinnings and Clinical Correlations. Semin Pediatr Neurol. 2020 Oct;35:100832. doi: 10.1016/j.spen.2020.100832. Epub 2020 Jun 24. PMID 32892959
- [Background] Barth B, Rohe T, Deppermann S, Fallgatter AJ, Ehlis AC. Neural oscillatory responses to performance monitoring differ between high- and low-impulsive individuals, but are unaffected by TMS. Hum Brain Mapp. 2021 Jun 1;42(8):2416-2433. doi: 10.1002/hbm.25376. Epub 2021 Feb 19. PMID 33605509